CLINICAL TRIAL: NCT05535283
Title: An Observational Study Investigating The Experiences of Patients In Osteosarcoma Clinical Trials
Brief Title: Assessing Clinical Trial Experiences of Patients With Osteosarcoma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83926159
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this study so that it may collect a variety of data about osteosarcoma clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with osteosarcoma who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with osteosarcoma
* Patient has self-identified as planning to enroll in an interventional clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* ECOG score of 4
* Patient is pregnant
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteosarcoma patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an osteosarcoma clinical trial | 3 months
Rate of patients who remain in osteosarcoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bielack S, Carrle D, Jost L; ESMO Guidelines Working Group. Osteosarcoma: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2008 May;19 Suppl 2:ii94-6. doi: 10.1093/annonc/mdn102. No abstract available. PMID 18456784
- [Background] Wittig JC, Bickels J, Priebat D, Jelinek J, Kellar-Graney K, Shmookler B, Malawer MM. Osteosarcoma: a multidisciplinary approach to diagnosis and treatment. Am Fam Physician. 2002 Mar 15;65(6):1123-32. PMID 11925089
- [Background] Burns L, Perisoglou M. Clinical trials in osteosarcoma treatment: patients' perspective through art. Recent Results Cancer Res. 2009;179:345-61. doi: 10.1007/978-3-540-77960-5_22. PMID 19230551

DOCUMENTS (1):
  • Informed Consent Form (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT05535283/ICF_000.pdf